CLINICAL TRIAL: NCT02853006
Title: Study on Fluids Associated to Lung Cancer, of the Ectopic Expression of Cancer Testis Gene and Mutation as Diagnostics and Prognosis Biomarkers
Brief Title: Study on Fluids Associated to Lung Cancer
Acronym: ECTOPIC/MUTAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 38RC15.099
Record Dates: First submitted 2016-07-13; First posted 2016-08-02 (Estimated); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Lung Cancer
Keywords: Cancer lung; Fluids; LungCancerTest; radiological anomalies; non-cancerous; carriers; Patient reference
MeSH Terms: conditions — Lung Neoplasms | interventions — Blood Specimen Collection; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 lung cancer in stage 1-2 (Other): Group 1 : patient with lung cancer in stage 1-2, lung cancer of all histology kind eligible for surgery
  Interventions: Biological: Blood and respiratory fluids sampling; Procedure: Excised tissues
- Group 2 lung cancer in stage 3-4 (Other): Group 2 : patient with lung cancer in stage 3-4 (no adenocarcinoma or squamous) receiving classical or targeted chemotherapy on genetic anomalies.
  Interventions: Biological: Blood and respiratory fluids sampling; Procedure: Biopsy
- Group 3 : control patients (Other): Group 3 control patients : carriers of non-cancerous radiological anomalies : benign nodules, cicatricial lesions, infectious or inflammatory, paired with the two other groups by age, sex or tobacco.
  Interventions: Biological: Blood and respiratory fluids sampling

INTERVENTIONS:
Biological: Blood and respiratory fluids sampling — In order to extract RNA (LungCancerTest) and DNA (mutation, reassortment).
Procedure: Biopsy
  Arms: Group 2 lung cancer in stage 3-4
Procedure: Excised tissues
  Arms: Group 1 lung cancer in stage 1-2

SUMMARY:
The diagnosis of lung cancer is the first cause of cancer deaths for man and woman. It requires invasive procedures (at least endoscopy, transthoracic puncture, or surgery).

This study is about the set up of an innovative test for lung cancer prognosis, based on biopsies and surgical material : LungCancerTest, with the creation of a start-up in progress.

The main goal of this study is to approve the diagnostic value of the molecular signature of the 26 genes (LungCancerTest) revealed in blood and respiratory fluids among patients with lung cancer.

ELIGIBILITY:
Inclusion Criterias :

* Patients with lung cancer in stage 1-2, lung cancer of all histology kind eligible for surgery (Group 1).
* Patients with lung cancer in stage 3-4 (no adenocarcinoma or squamous) receiving classical or targeted chemotherapy on genetic anomalies (Group 2).
* Control patients : carriers of non-cancerous radiological anomalies : benign nodules, cicatricial lesions, infectious or inflammatory, paired with the two other groups by age, sex or tobacco (Group 3).
* Adults patients : over 18 years.
* Persons affiliated to national social security.
* Free signed consent.

Exclusion Criterias :

* Persons referred to in articles L1121-5 to L1121-8 of CSP ( protected people) : pregnants, parturients or breastfeeding women, person deprived of liberty by judicial or administrative decision, person under legal protection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2015-06; Primary Completion 2019-09 (Actual); Study Completion 2020-02 (Actual)

PRIMARY OUTCOMES:
Quantification of : DNA | Half a day
  From plasma or respiratory fluids, with Qiagen QIAamp MinElute Virus Spin kit.
  Picogreen technique (fluorimétrie) with the device Qubit 2.0 Characterization of DNA by migration on revealed agarose gel in presence of ethidium bromide
  Study of DNA (mutation, reassortment) with New Generation Sequencing materiel.
Quantification of : RNA | Half a day
  From plasma or respiratory fluids, with Qiagen QIAamp MinElute Virus Spin kit.
  Picogreen technique (fluorimétrie) with the device Qubit 2.0 Characterization of RNA with an Agilent chip
  Study of RNA (LungCancerTest) with PCR-Array prototype to show the expression of the molecular signature (Cancer Testis genes).

CONTACTS AND LOCATIONS:
Overall Officials: Christian Brambilla, Professor, Principal Investigator — Grenoble Hospital University
Locations (1):
- UniversityHospitalGrenoble, La Tronche, France

REFERENCES:
- [Background] Toffart AC, Timsit JF, Couraud S, Merle P, Moro-Sibilot D, Perol M, Mastroianni B, Souquet PJ, Girard N, Jeannin G, Romand P, Chatellain P, Vesin A, Brambilla C, Brambilla E. Immunohistochemistry evaluation of biomarker expression in non-small cell lung cancer (Pharmacogenoscan study). Lung Cancer. 2014 Feb;83(2):182-8. doi: 10.1016/j.lungcan.2013.12.003. Epub 2013 Dec 21. PMID 24388706
- [Background] Rousseaux S, Debernardi A, Jacquiau B, Vitte AL, Vesin A, Nagy-Mignotte H, Moro-Sibilot D, Brichon PY, Lantuejoul S, Hainaut P, Laffaire J, de Reynies A, Beer DG, Timsit JF, Brambilla C, Brambilla E, Khochbin S. Ectopic activation of germline and placental genes identifies aggressive metastasis-prone lung cancers. Sci Transl Med. 2013 May 22;5(186):186ra66. doi: 10.1126/scitranslmed.3005723. PMID 23698379
- [Background] BRAMBILLA C., ROUSSEAUX S., DE BERNARDI A., JACQUIAU B., VITTE A.L., ARBIB F., LEMAITRE N., LANTUEJOUL S., MIGNOTTE H, MORO-SIBILOT D., TOFFART A.C., BRAMBILLA E., KOCHBIN S. A PCR-based test detecting ectopic expressions of placenta/germline genes can predict aggressive lung tumours. J. Thor. Oncol. • Volume 8, Supplement 2, November 2013 S1048
- [Background] Vignot S, Frampton GM, Soria JC, Yelensky R, Commo F, Brambilla C, Palmer G, Moro-Sibilot D, Ross JS, Cronin MT, Andre F, Stephens PJ, Lazar V, Miller VA, Brambilla E. Next-generation sequencing reveals high concordance of recurrent somatic alterations between primary tumor and metastases from patients with non-small-cell lung cancer. J Clin Oncol. 2013 Jun 10;31(17):2167-72. doi: 10.1200/JCO.2012.47.7737. Epub 2013 Apr 29. PMID 23630207
- [Background] PEIFER M, FERNÁNDEZ-CUESTA L, SOS ML, GEORGE J, SEIDEL D, KASPER LH, PLENKER D, LEENDERS F, SUN R, ZANDER T, MENON R, KOKER M, DAHMEN I, MÜLLER C, DI CERBO V, SCHILDHAUS HU, ALTMÜLLER J, BAESSMANN I, BECKER C, DE WILDE B, VANDESOMPELE J, BÖHM D, ANSÉN S, GABLER F, WILKENING I, HEYNCK S, HEUCKMANN JM, LU X, CARTER SL, CIBULSKIS K, BANERJI S, GETZ G, PARK KS, RAUH D, GRÜTTER C, FISCHER M, PASQUALUCCI L, WRIGHT G, WAINER Z, RUSSELL P, PETERSEN I, CHEN Y, STOELBEN E, LUDWIG C, SCHNABEL P, HOFFMANN H, MULEY T, BROCKMANN M, ENGEL-RIEDEL W, MUSCARELLA LA, FAZIO VM, GROEN H, TIMENS W, SIETSMA H, THUNNISSEN E, SMIT E, HEIDEMAN DA, SNIJDERS PJ, CAPPUZZO F, LIGORIO C, DAMIANI S, FIELD J, SOLBERG S, BRUSTUGUN OT, LUND-IVERSEN M, SÄNGER J, CLEMENT JH, SOLTERMANN A, MOCH H, WEDER W, SOLOMON B, SORIA JC, VALIDIRE P, BESSE B, BRAMBILLA E, BRAMBILLA C, LANTUEJOUL S, LORIMIER P, SCHNEIDER PM, HALLEK M, PAO W, MEYERSON M, SAGE J, SHENDURE J, SCHNEIDER R, BÜTTNER R, WOLF J, NÜRNBERG P, PERNER S, HEUKAMP LC, BRINDLE PK, HAAS S, THOMAS RK. Integrative genome analyses identify key somatic driver mutations of small-cell lung cancer.Nat Genet. 2012;44(10):1104-10
- [Background] Nagy-Mignotte H, Guillem P, Vignoud L, Coudurier M, Vesin A, Bonneterre V, Toffart AC, Sakhri L, Brambilla C, Brambilla E, Timsit JF, Moro-Sibilot D; Multidisciplinary Thoracic Oncology Group. Outcomes in recurrent small-cell lung cancer after one to four chemotherapy lines: a retrospective study of 300 patients. Lung Cancer. 2012 Oct;78(1):112-20. doi: 10.1016/j.lungcan.2012.06.006. Epub 2012 Jul 12. PMID 22795703
- [Background] Lecourtois B, Jankowski A, Arbib F, Lantuejoul S, Brichon PY, Moro-Sibilot D, Brambilla C, Ferretti G. Endobronchial tumours in a campaign for early detection of bronchial cancer: Computed tomography versus endoscopy. Diagn Interv Imaging. 2012 Jul;93(7-8):604-11. doi: 10.1016/j.diii.2012.05.002. Epub 2012 Jul 6. PMID 22771372
- [Background] Mortamais M, Chevrier C, Philippat C, Petit C, Calafat AM, Ye X, Silva MJ, Brambilla C, Eijkemans MJ, Charles MA, Cordier S, Slama R. Correcting for the influence of sampling conditions on biomarkers of exposure to phenols and phthalates: a 2-step standardization method based on regression residuals. Environ Health. 2012 Apr 26;11:29. doi: 10.1186/1476-069X-11-29. PMID 22537080
- [Background] Brambilla C, Sanchez-Chardi A, Perez-Trujillo M, Julian E, Luquin M. Cyclopropanation of alpha-mycolic acids is not required for cording in Mycobacterium brumae and Mycobacterium fallax. Microbiology (Reading). 2012 Jun;158(Pt 6):1615-1621. doi: 10.1099/mic.0.057919-0. Epub 2012 Apr 5. PMID 22493302
- [Background] Han N, Dol Z, Vasieva O, Hyde R, Liloglou T, Raji O, Brambilla E, Brambilla C, Martinet Y, Sozzi G, Risch A, Montuenga LM; EUELC Consortium; Brass A, Field JK. Progressive lung cancer determined by expression profiling and transcriptional regulation. Int J Oncol. 2012 Jul;41(1):242-52. doi: 10.3892/ijo.2012.1421. Epub 2012 Mar 28. PMID 22469662
- [Background] Pajares MJ, Agorreta J, Larrayoz M, Vesin A, Ezponda T, Zudaire I, Torre W, Lozano MD, Brambilla E, Brambilla C, Wistuba II, Behrens C, Timsit JF, Pio R, Field JK, Montuenga LM. Expression of tumor-derived vascular endothelial growth factor and its receptors is associated with outcome in early squamous cell carcinoma of the lung. J Clin Oncol. 2012 Apr 1;30(10):1129-36. doi: 10.1200/JCO.2011.37.4231. Epub 2012 Feb 21. PMID 22355056
- [Background] Hammerman PS, Sos ML, Ramos AH, Xu C, Dutt A, Zhou W, Brace LE, Woods BA, Lin W, Zhang J, Deng X, Lim SM, Heynck S, Peifer M, Simard JR, Lawrence MS, Onofrio RC, Salvesen HB, Seidel D, Zander T, Heuckmann JM, Soltermann A, Moch H, Koker M, Leenders F, Gabler F, Querings S, Ansen S, Brambilla E, Brambilla C, Lorimier P, Brustugun OT, Helland A, Petersen I, Clement JH, Groen H, Timens W, Sietsma H, Stoelben E, Wolf J, Beer DG, Tsao MS, Hanna M, Hatton C, Eck MJ, Janne PA, Johnson BE, Winckler W, Greulich H, Bass AJ, Cho J, Rauh D, Gray NS, Wong KK, Haura EB, Thomas RK, Meyerson M. Mutations in the DDR2 kinase gene identify a novel therapeutic target in squamous cell lung cancer. Cancer Discov. 2011 Jun;1(1):78-89. doi: 10.1158/2159-8274.CD-11-0005. PMID 22328973
- [Background] Scoccianti C, Vesin A, Martel G, Olivier M, Brambilla E, Timsit JF, Tavecchio L, Brambilla C, Field JK, Hainaut P; European Early Lung Cancer Consortium. Prognostic value of TP53, KRAS and EGFR mutations in nonsmall cell lung cancer: the EUELC cohort. Eur Respir J. 2012 Jul;40(1):177-84. doi: 10.1183/09031936.00097311. Epub 2012 Jan 20. PMID 22267755
- [Background] Philippat C, Mortamais M, Chevrier C, Petit C, Calafat AM, Ye X, Silva MJ, Brambilla C, Pin I, Charles MA, Cordier S, Slama R. Exposure to phthalates and phenols during pregnancy and offspring size at birth. Environ Health Perspect. 2012 Mar;120(3):464-70. doi: 10.1289/ehp.1103634. Epub 2011 Sep 7. PMID 21900077
- [Background] Thunnissen FB, Prinsen C, Hol B, Van der Drift M, Vesin A, Brambilla C, Montuenga L, Field JK; EUELC consortium. Smoking history and lung carcinoma: KRAS mutation is an early hit in lung adenocarcinoma development. Lung Cancer. 2012 Feb;75(2):156-60. doi: 10.1016/j.lungcan.2011.07.013. Epub 2011 Aug 11. PMID 21839537
- [Background] Nagy-Mignotte H, Guillem P, Vesin A, Toffart AC, Colonna M, Bonneterre V, Brichon PY, Brambilla C, Brambilla E, Lantuejoul S, Timsit JF, Moro-Sibilot D; Multidisciplinary Thoracic Oncology Group at Grenoble University Hospital. Primary lung adenocarcinoma: characteristics by smoking habit and sex. Eur Respir J. 2011 Dec;38(6):1412-9. doi: 10.1183/09031936.00191710. Epub 2011 Aug 4. PMID 21828037
- [Background] Bousquet J, Anto JM, Sterk PJ, Adcock IM, Chung KF, Roca J, Agusti A, Brightling C, Cambon-Thomsen A, Cesario A, Abdelhak S, Antonarakis SE, Avignon A, Ballabio A, Baraldi E, Baranov A, Bieber T, Bockaert J, Brahmachari S, Brambilla C, Bringer J, Dauzat M, Ernberg I, Fabbri L, Froguel P, Galas D, Gojobori T, Hunter P, Jorgensen C, Kauffmann F, Kourilsky P, Kowalski ML, Lancet D, Pen CL, Mallet J, Mayosi B, Mercier J, Metspalu A, Nadeau JH, Ninot G, Noble D, Ozturk M, Palkonen S, Prefaut C, Rabe K, Renard E, Roberts RG, Samolinski B, Schunemann HJ, Simon HU, Soares MB, Superti-Furga G, Tegner J, Verjovski-Almeida S, Wellstead P, Wolkenhauer O, Wouters E, Balling R, Brookes AJ, Charron D, Pison C, Chen Z, Hood L, Auffray C. Systems medicine and integrated care to combat chronic noncommunicable diseases. Genome Med. 2011 Jul 6;3(7):43. doi: 10.1186/gm259. PMID 21745417
- [Background] Edmond V, Brambilla C, Brambilla E, Gazzeri S, Eymin B. SRSF2 is required for sodium butyrate-mediated p21(WAF1) induction and premature senescence in human lung carcinoma cell lines. Cell Cycle. 2011 Jun 15;10(12):1968-77. doi: 10.4161/cc.10.12.15825. Epub 2011 Jun 15. PMID 21555914
- [Background] Travis WD, Brambilla E, Noguchi M, Nicholson AG, Geisinger KR, Yatabe Y, Beer DG, Powell CA, Riely GJ, Van Schil PE, Garg K, Austin JH, Asamura H, Rusch VW, Hirsch FR, Scagliotti G, Mitsudomi T, Huber RM, Ishikawa Y, Jett J, Sanchez-Cespedes M, Sculier JP, Takahashi T, Tsuboi M, Vansteenkiste J, Wistuba I, Yang PC, Aberle D, Brambilla C, Flieder D, Franklin W, Gazdar A, Gould M, Hasleton P, Henderson D, Johnson B, Johnson D, Kerr K, Kuriyama K, Lee JS, Miller VA, Petersen I, Roggli V, Rosell R, Saijo N, Thunnissen E, Tsao M, Yankelewitz D. International association for the study of lung cancer/american thoracic society/european respiratory society international multidisciplinary classification of lung adenocarcinoma. J Thorac Oncol. 2011 Feb;6(2):244-85. doi: 10.1097/JTO.0b013e318206a221. PMID 21252716
- [Background] Garelli M, Righini C, Faure C, Jankowski A, Brambilla C, Ferretti GR. Imaging of a case of extramedullary solitary plasmacytoma of the trachea. Case Rep Radiol. 2011;2011:687203. doi: 10.1155/2011/687203. Epub 2011 Sep 22. PMID 22606554
- [Background] Weiss J, Sos ML, Seidel D, Peifer M, Zander T, Heuckmann JM, Ullrich RT, Menon R, Maier S, Soltermann A, Moch H, Wagener P, Fischer F, Heynck S, Koker M, Schottle J, Leenders F, Gabler F, Dabow I, Querings S, Heukamp LC, Balke-Want H, Ansen S, Rauh D, Baessmann I, Altmuller J, Wainer Z, Conron M, Wright G, Russell P, Solomon B, Brambilla E, Brambilla C, Lorimier P, Sollberg S, Brustugun OT, Engel-Riedel W, Ludwig C, Petersen I, Sanger J, Clement J, Groen H, Timens W, Sietsma H, Thunnissen E, Smit E, Heideman D, Cappuzzo F, Ligorio C, Damiani S, Hallek M, Beroukhim R, Pao W, Klebl B, Baumann M, Buettner R, Ernestus K, Stoelben E, Wolf J, Nurnberg P, Perner S, Thomas RK. Frequent and focal FGFR1 amplification associates with therapeutically tractable FGFR1 dependency in squamous cell lung cancer. Sci Transl Med. 2010 Dec 15;2(62):62ra93. doi: 10.1126/scitranslmed.3001451. PMID 21160078
- [Background] Edmond V, Moysan E, Khochbin S, Matthias P, Brambilla C, Brambilla E, Gazzeri S, Eymin B. Acetylation and phosphorylation of SRSF2 control cell fate decision in response to cisplatin. EMBO J. 2011 Feb 2;30(3):510-23. doi: 10.1038/emboj.2010.333. Epub 2010 Dec 14. PMID 21157427
- [Background] Larrieu D, Ythier D, Brambilla C, Pedeux R. ING2 controls the G1 to S-phase transition by regulating p21 expression. Cell Cycle. 2010 Oct 1;9(19):3984-90. doi: 10.4161/cc.9.19.13208. Epub 2010 Oct 1. PMID 20890119
- [Background] Ythier D, Larrieu D, Binet R, Binda O, Brambilla C, Gazzeri S, Pedeux R. Sumoylation of ING2 regulates the transcription mediated by Sin3A. Oncogene. 2010 Nov 4;29(44):5946-56. doi: 10.1038/onc.2010.325. Epub 2010 Aug 2. PMID 20676127
- [Background] Bryant CM, Albertus DL, Kim S, Chen G, Brambilla C, Guedj M, Arima C, Travis WD, Yatabe Y, Takahashi T, Brambilla E, Beer DG. Clinically relevant characterization of lung adenocarcinoma subtypes based on cellular pathways: an international validation study. PLoS One. 2010 Jul 22;5(7):e11712. doi: 10.1371/journal.pone.0011712. PMID 20661423
- [Background] Merdzhanova G, Gout S, Keramidas M, Edmond V, Coll JL, Brambilla C, Brambilla E, Gazzeri S, Eymin B. The transcription factor E2F1 and the SR protein SC35 control the ratio of pro-angiogenic versus antiangiogenic isoforms of vascular endothelial growth factor-A to inhibit neovascularization in vivo. Oncogene. 2010 Sep 30;29(39):5392-403. doi: 10.1038/onc.2010.281. Epub 2010 Jul 19. PMID 20639906
- [Background] Van den Berg RM, Brokx H, Vesin A, Field JK, Brambilla C, Meijer CJ, Sutedja GT, Heideman DA, Postmus PE, Smit EF, Snijders PJ. Prognostic value of hTERT mRNA expression in surgical samples of lung cancer patients: the European Early Lung Cancer Project. Int J Oncol. 2010 Aug;37(2):455-61. doi: 10.3892/ijo_00000694. PMID 20596673
- [Background] Caron C, Lestrat C, Marsal S, Escoffier E, Curtet S, Virolle V, Barbry P, Debernardi A, Brambilla C, Brambilla E, Rousseaux S, Khochbin S. Functional characterization of ATAD2 as a new cancer/testis factor and a predictor of poor prognosis in breast and lung cancers. Oncogene. 2010 Sep 16;29(37):5171-81. doi: 10.1038/onc.2010.259. Epub 2010 Jun 28. PMID 20581866
- [Background] Lantuejoul S, Raynaud C, Salameire D, Gazzeri S, Moro-Sibilot D, Soria JC, Brambilla C, Brambilla E. Telomere maintenance and DNA damage responses during lung carcinogenesis. Clin Cancer Res. 2010 Jun 1;16(11):2979-88. doi: 10.1158/1078-0432.CCR-10-0142. Epub 2010 Apr 19. PMID 20404006
- [Background] Ythier D, Brambilla E, Binet R, Nissou D, Vesin A, de Fraipont F, Moro-Sibilot D, Lantuejoul S, Brambilla C, Gazzeri S, Pedeux R. Expression of candidate tumor suppressor gene ING2 is lost in non-small cell lung carcinoma. Lung Cancer. 2010 Aug;69(2):180-6. doi: 10.1016/j.lungcan.2009.11.006. Epub 2009 Dec 4. PMID 19962781
- [Background] Wattrelot P, Brion JP, Labarere J, Billette de Villemeur A, Girard-Blanc MF, Stahl JP, Brambilla C. [Vaccination practices following the end of compulsory BCG vaccination. A cross-sectional survey of general practitioners and pediatricians]. Arch Pediatr. 2010 Feb;17(2):118-24. doi: 10.1016/j.arcped.2009.10.025. Epub 2009 Dec 2. French. PMID 19959346
- [Background] Binet R, Ythier D, Robles AI, Collado M, Larrieu D, Fonti C, Brambilla E, Brambilla C, Serrano M, Harris CC, Pedeux R. WNT16B is a new marker of cellular senescence that regulates p53 activity and the phosphoinositide 3-kinase/AKT pathway. Cancer Res. 2009 Dec 15;69(24):9183-91. doi: 10.1158/0008-5472.CAN-09-1016. PMID 19951988
- [Background] Field JK, Liloglou T, Niaz A, Bryan J, Gosney JR, Giles T, Brambilla C, Brambilla E, Vesin A, Timsit JF, Hainaut P, Martinet Y, Vignaud JM, Thunnissen FB, Prinsen C, Snijders PJ, Smit EF, Sozzi G, Roz L, Risch A, Becker HD, Elborn JS, Magee ND, Montuenga LM, Pajares MJ, Lozano MD, O'Byrne KJ, Harrison DJ, Niklinski J, Cassidy A; EUELC Collaborators. EUELC project: a multi-centre, multipurpose study to investigate early stage NSCLC, and to establish a biobank for ongoing collaboration. Eur Respir J. 2009 Dec;34(6):1477-86. doi: 10.1183/09031936.00077809. PMID 19948914
- [Background] Felix L, Serra-Tosio G, Lantuejoul S, Timsit JF, Moro-Sibilot D, Brambilla C, Ferretti GR. CT characteristics of resolving ground-glass opacities in a lung cancer screening programme. Eur J Radiol. 2011 Mar;77(3):410-6. doi: 10.1016/j.ejrad.2009.09.008. Epub 2009 Oct 4. PMID 19804950
- [Background] Larrieu D, Ythier D, Binet R, Brambilla C, Brambilla E, Sengupta S, Pedeux R. ING2 controls the progression of DNA replication forks to maintain genome stability. EMBO Rep. 2009 Oct;10(10):1168-74. doi: 10.1038/embor.2009.180. Epub 2009 Sep 4. PMID 19730436
- [Background] Cassidy A, Balsan J, Vesin A, Wu X, Liloglou T, Brambilla C, Timsit JF, Field JK; EUELC Consortium. Cancer diagnosis in first-degree relatives and non-small cell lung cancer risk: results from a multi-centre case-control study in Europe. Eur J Cancer. 2009 Nov;45(17):3047-53. doi: 10.1016/j.ejca.2009.05.006. Epub 2009 May 29. PMID 19482469
- [Background] Delloye-Bourgeois C, Brambilla E, Coissieux MM, Guenebeaud C, Pedeux R, Firlej V, Cabon F, Brambilla C, Mehlen P, Bernet A. Interference with netrin-1 and tumor cell death in non-small cell lung cancer. J Natl Cancer Inst. 2009 Feb 18;101(4):237-47. doi: 10.1093/jnci/djn491. Epub 2009 Feb 10. PMID 19211441
- [Background] Brambilla C. From surgical to molecular scalpel: ERJ lung cancer series for 2009. Eur Respir J. 2009 Jan;33(1):9-10. doi: 10.1183/09031936.00162908. No abstract available. PMID 19123267
- [Background] Verri C, Roz L, Conte D, Liloglou T, Livio A, Vesin A, Fabbri A, Andriani F, Brambilla C, Tavecchio L, Calarco G, Calabro E, Mancini A, Tosi D, Bossi P, Field JK, Brambilla E, Sozzi G; EUELC Consortium. Fragile histidine triad gene inactivation in lung cancer: the European Early Lung Cancer project. Am J Respir Crit Care Med. 2009 Mar 1;179(5):396-401. doi: 10.1164/rccm.200807-1153OC. Epub 2008 Dec 18. PMID 19096006
- [Background] Van Den Broeck A, Brambilla E, Moro-Sibilot D, Lantuejoul S, Brambilla C, Eymin B, Gazzeri S. Loss of histone H4K20 trimethylation occurs in preneoplasia and influences prognosis of non-small cell lung cancer. Clin Cancer Res. 2008 Nov 15;14(22):7237-45. doi: 10.1158/1078-0432.CCR-08-0869. Epub 2008 Oct 30. PMID 18974389
- [Background] Merdzhanova G, Edmond V, De Seranno S, Van den Broeck A, Corcos L, Brambilla C, Brambilla E, Gazzeri S, Eymin B. E2F1 controls alternative splicing pattern of genes involved in apoptosis through upregulation of the splicing factor SC35. Cell Death Differ. 2008 Dec;15(12):1815-23. doi: 10.1038/cdd.2008.135. Epub 2008 Sep 19. PMID 18806759
- [Background] Ythier D, Larrieu D, Brambilla C, Brambilla E, Pedeux R. The new tumor suppressor genes ING: genomic structure and status in cancer. Int J Cancer. 2008 Oct 1;123(7):1483-90. doi: 10.1002/ijc.23790. PMID 18636562
- [Background] Bertrand D, Righini C, Ferretti G, Brambilla C, Moro-Sibilot D. [Early diagnosis of bronchial carcinoma after head and neck cancer]. Rev Mal Respir. 2008 May;25(5):559-68. doi: 10.1016/s0761-8425(08)71613-9. French. PMID 18535523
- [Background] Ferretti GR, Jankowski A, Rodiere M, Brichon PY, Brambilla C, Lantuejoul S. CT-guided biopsy of nonresolving focal air space consolidation. J Thorac Imaging. 2008 Feb;23(1):7-12. doi: 10.1097/RTI.0b013e3181453e04. PMID 18347513
- [Background] Brambilla C, Colonna M. Cannabis: the next villain on the lung cancer battlefield? Eur Respir J. 2008 Feb;31(2):227-8. doi: 10.1183/09031936.00157607. No abstract available. PMID 18238942